CLINICAL TRIAL: NCT02355574
Title: An Ongoing, 5-year Post Market Study to Track Clinical Application of DecisionDx-Melanoma Gene Expression Profile (GEP) Assay Results and the Impact on Patient Outcomes and Health Economics
Brief Title: 5-year Study to Track Clinical Application of DecisionDx-Melanoma Gene Expression Profile Assay Results
Acronym: INTEGRATE
Status: Terminated | Type: Observational
Why Stopped: Study endpoints completed with lower than anticipated enrollment. Last patient enrolled completed final visit February 2021.
Sponsor: Castle Biosciences Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: INTEGRATE_1_Protocol
Record Dates: First submitted 2014-12-18; First posted 2015-02-04 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Cutaneous Melanoma
Keywords: melanoma; cutaneous melanoma; DecisionDx-Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The INTEGRATE Registry Study follows patients with cutaneous melanoma who have had the DecisionDx-Melanoma gene expression assay performed. Data will be collected through review of medical records from clinical visits with physician.

The purpose is to document the clinical application of results obtained from the DecisionDx- Melanoma multi-gene assay and to track outcomes of patients for whom DecisionDx-Melanoma testing has been completed. Additionally the study will assess the health economic impact of DecisionDx-Melanoma testing as it relates to the Melanoma population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with melanoma and determined, by their physician, to be appropriate for DecisionDx-Melanoma testing and who have successful results available to the investigator are eligible for registration
* Patients enrolled should be reasonably able to follow-up with the enrolling physician at regular intervals for assessment of outcome data.
* 16 Years and older

Exclusion Criteria:

* Less than 16 Years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cutaneous melanoma for whom DecisionDx-Melanoma testing is to be clinically performed.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Adjusted surveillance regimen | upon receipt DecisionDX-Melanoma results received and every 6 months thereafter
  * Relaxed surveillance for the low risk group;
  * Increased vigilance for early detection in the high risk group.

SECONDARY OUTCOMES:
Referral for sentinel lymph node interrogation in the high risk group in thin melanomas. | Upon receipt DecisionDx-Melanoma results
  referral to SLNB in HR melanoma

OTHER OUTCOMES:
Early referral to medical oncologist for high risk patients. | Upon Receipt DecisionDx-Melanoma results
  referral

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cook, PhD, Principal Investigator — Castle Biosciences Inc.
Locations (3):
- United States (3):
  - Northside Hospital, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Saint Louis University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitman ED, Koshenkov VP, Gastman BR, Lewis D, Hsueh EC, Pak H, Trezona TP, Davidson RS, McPhee M, Guenther JM, Toomey P, Smith FO, Beitsch PD, Lewis JM, Ward A, Young SE, Shah PK, Quick AP, Martin BJ, Zolochevska O, Covington KR, Monzon FA, Goldberg MS, Cook RW, Fleming MD, Hyams DM, Vetto JT. Integrating 31-Gene Expression Profiling With Clinicopathologic Features to Optimize Cutaneous Melanoma Sentinel Lymph Node Metastasis Prediction. JCO Precis Oncol. 2021 Sep 13;5:PO.21.00162. doi: 10.1200/PO.21.00162. eCollection 2021. PMID 34568719
- [Derived] Hsueh EC, DeBloom JR, Lee JH, Sussman JJ, Covington KR, Caruso HG, Quick AP, Cook RW, Slingluff CL Jr, McMasters KM. Long-Term Outcomes in a Multicenter, Prospective Cohort Evaluating the Prognostic 31-Gene Expression Profile for Cutaneous Melanoma. JCO Precis Oncol. 2021 Apr 6;5:PO.20.00119. doi: 10.1200/PO.20.00119. eCollection 2021. PMID 34036233